CLINICAL TRIAL: NCT04190654
Title: A Pharmacokinetic Study of KW-6356 in Subjects With Mild and Moderate Hepatic Impairment Compared to Subjects With Normal Hepatic Function
Brief Title: Single-dose Study to Investigate the Plasma PK of KW-6356 and Its Major Metabolite
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Kyowa Kirin, Inc. (Industry)
Responsible Party: Sponsor
Organization: Kyowa Kirin Co., Ltd. (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 6356-006
Record Dates: First submitted 2019-11-25; First posted 2019-12-09 (Actual); Last update posted 2024-04-25 (Actual); Status verified 2024-04

CONDITIONS: Hepatic Impairment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Mild Hepatic Impairment (Experimental): Subjects with mild hepatic impairment (Child-Pugh class A score of 5 or 6)
  Interventions: Drug: KW-6356
- Moderate Hepatic Impairment (Experimental): Subjects with moderate hepatic impairment (Child-Pugh class B score of 7 to 9)
  Interventions: Drug: KW-6356
- Healthy Subjects (Experimental): Healthy adults matched with the subjects in Group A and Group B at 1:1 for age (± 10 years), sex, and BMI (± 20%)
  Interventions: Drug: KW-6356

INTERVENTIONS:
Drug: KW-6356 — Single oral dose of KW-6356

SUMMARY:
This is an open-label, non-randomized, single-dose study to investigate the plasma PK of KW-6356 and its major metabolite, after a single oral dose of KW-6356, in subjects with mild or moderate hepatic impairment and in healthy adults

DETAILED DESCRIPTION:
Potential subjects will be screened to assess their eligibility to enter the study within 4 weeks prior to dose administration. Eligible subjects will be admitted to the clinical research unit (CRU) before the initiation of investigational medicinal product (IMP) administration (Check-in/Day -1) and administered of KW-6356 orally on Day 1 after an 8-hour fast. Those subjects who complete all the scheduled observations/examinations and are determined to have no clinical abnormalities requiring further hospitalization by the Investigator, will be discharged from the study site on Day 4. Discharged subjects will then visit the CRU on the scheduled visit Days 5, 6, 7, 8 for PK sample collections and safety assessments on Day 12 to complete the End of Study (EOS) visit. The duration of hospitalization will be 5 days: 4 nights from Day -1 to Day 4.

ELIGIBILITY:
Inclusion Criteria:

All Subjects:

1. Individuals who provide freely given written consent for participating in the study.
2. Men and women aged ≥ 18 and ≤ 75 years at the date of providing informed consent.
3. Subjects with a BMI in the range 18.0 to 40.0 kg/m2.
4. Females will not be pregnant or lactating, and females of childbearing potential and males will agree to use contraception.
5. Able to comprehend and willing to sign an ICF and to abide by the study restrictions.

   Subjects with Hepatic Impairment:
6. Subjects must meet the criteria for mild or moderate hepatic impairment based on CP classification. Subjects will be classified at Screening based on CP score and classification will be repeated at Check-in. If the hepatic function classification for the subject is not the same at the 2 timepoints, enrollment of the subject into a hepatic category group will be based on the CP score at Screening.
7. Subjects have stable hepatic function with a diagnosis of chronic disease of > 6 months, defined as no clinically significant change in disease status within the 60 days prior to the Screening visit or 90 days prior to drug administration on Day 1 (whichever is longer), as documented by the subject's recent medical history.
8. Subjects are on a stable medication dose(s) and/or treatment regimen(s) for treatment of hepatic impairment during the 30 days preceding the first dose of IMP. Drugs known to be moderate-to-potent inhibitors or inducers of CYP3A4/5 enzyme will not be allowed. Subjects requiring medications that are moderate-to-potent inhibitors or inducers of CYP3A4/5 may have these medications discontinued for purposes of qualifying for at least 30 days prior to dosing day for this study. Adjustments may be made if deemed medically safe and also acceptable to the Sponsor and Medical Monitor.
9. Subjects with mild or moderate hepatic impairment may have medical findings consistent with their hepatic dysfunction, as determined by medical history, physical examination, 12-lead ECG, vital sign measurements, and clinical laboratory evaluations at Screening and Check-in. Subjects with abnormal findings considered not clinically significant by the Investigator will be eligible. Vital signs between the following ranges and stable (measured in a supine position after a minimum of 5 minutes supine):

   1. Systolic blood pressure ≥ 90 and ≤ 160 mmHg
   2. Diastolic blood pressure ≥ 50 and ≤ 95 mmHg
   3. Pulse rate ≥ 45 and ≤ 100 bpm

   Healthy Subjects with Normal Hepatic Function:
10. Subjects with no clinically significant abnormalities in liver function test results (AST, ALT, gamma-glutamyl transferase [γ-GTP], alkaline phosphatase, total bilirubin, albumin [Alb], and PT) at Screening and Check-in. In good health, determined by no clinically significant findings from medical history, physical examination, 12-lead ECG, vital signs measurements, and clinical laboratory evaluations (congenital nonhemolytic hyperbilirubinemia [eg, suspicion of Gilbert's syndrome based on total and direct bilirubin] is not acceptable) at Screening and Check-in as assessed by the Investigator. Vital signs between the following ranges and stable (measured in a supine position after a minimum of 5 minutes supine):

    1. Systolic blood pressure ≥ 95 and ≤ 150 mmHg mmHg
    2. Diastolic blood pressure ≥ 50 and ≤ 90 mmHg
    3. Pulse rate ≥ 45 and ≤ 100 bpm

Exclusion Criteria:

All Subjects:

1. Significant history or clinical manifestation of any metabolic, allergic, dermatological, renal, hematological, pulmonary, cardiovascular, gastrointestinal, neurological, respiratory, endocrine, or clinically significant psychiatric disorder, as determined by the Investigator. History of significant hypersensitivity, intolerance, or allergy to any drug compound, food, or other substance, unless approved by the Investigator.
2. History of stomach or intestinal surgery or resection that would potentially alter absorption and/or excretion of orally administered drugs (uncomplicated appendectomy, hernia repair, and cholecystectomy will be allowed).
3. Use of any prescriptions or substances that are known to be moderate to strong inducers or inhibitors of CYP3A4/5 within 30 days prior to dosing and during the study.
4. Use or intend to use any medications/products known to alter drug absorption, metabolism, or elimination processes, including St. John's wort, within 30 days prior to dosing, unless deemed acceptable by the Investigator.
5. Consumption of foods and beverages containing poppy seeds, grapefruit, or Seville oranges from 7 days prior to dosing until End of Study.
6. Consumption of caffeine-containing foods and beverages from 48 hours prior to Check-in.
7. Poor peripheral venous access.
8. Engaged in strenuous exercise within 7 days of Check-in.
9. Alcohol consumption is prohibited from 72 hours prior to dosing and during the study.
10. Subjects who were dosed in another clinical trial, or equivalent study of a drug or medical device, within 30 days, or 5 times the half-life of the IMP (whichever is longer) prior to IMP administration in the current study.
11. Subjects with receipt of blood products within 2 months prior to Check-in.
12. Subjects with donation of blood (> 200 mL) from 3 months prior to Screening, donation of plasma from 2 weeks prior to Screening, or donation of platelets from 6 weeks prior to Screening.
13. Subjects who test positive for acquired human immunodeficiency virus, including positive serology test results for hepatitis B surface antigen and/or human immunodeficiency virus 1/2. Subjects whose results are compatible with prior immunization for hepatitis B or natural immunity, and who tested positive for isolated hepatitis B core antibody with viral load negative may be included at the discretion of the Investigator.
14. Subjects who test positive for drugs of abuse at Screening and Check-in, with the exception of prescribed opioids and tetrahydrocannabinols (THC, marijuana) for pain management (Investigator verification required).
15. Subjects with positive urine drug screen for drugs of abuse at Screening and Check-in (opiates, amphetamines, methamphetamines, cannabinoids, benzodiazepines, cocaine, barbiturates, or methadone) or positive alcohol test (at Check-in only). Additionally, subjects who test positive for benzodiazepines may be allowed if prescribed under the care of a physician and reviewed/verified by Investigator.
16. Subjects with suicidal ideation or a positive score on the Baseline Columbia-Suicide Severity Rating Scale (C-SSRS).
17. Subjects with current or a history of significant hypersensitivity, intolerance, or allergy to any drug compound, food, or other substance, unless approved by the Investigator.
18. Subjects who contracted an infectious disease requiring hospitalization within 8 weeks prior to Screening.
19. Subjects who have previously received KW-6356.
20. Any other subjects who are determined by the Principal Investigator to be unsuitable for participation in this study.
21. Subjects with any current disease requiring treatment making study participation difficult, as determined by the Principal Investigator. Specifically, subjects with cardiovascular, clinically significant psychiatric, or gastrointestinal disorders are excluded.

    Subjects with Hepatic Impairment:
22. Subject smokes more than 10 cigarettes (ie, 1/2 pack) per day or equivalent (eg, e-vapor cigarette, pipe, cigar, chewing tobacco, nicotine patch, nicotine gum) and is unable to abstain from the use of tobacco products within 2 hours prior to and 4 hours after dose administration.
23. Subject has an alpha-fetoprotein level > 50 ng/mL.
24. History of paracentesis within 3 months prior to Check-in. Subject has required new medication for hepatic encephalopathy or an increase in dose of present medication for hepatic encephalopathy within 3 months prior to Check-in.
25. Subject has used prescription drugs within 14 days of IMP administration, with the exception of established therapy for hepatic disease and the treatment of disorders that have been stable for at least 30 days before IMP administration, as approved by the Investigator and in consultation with the Sponsor's Medical Monitor.
26. History of drug abuse within 1 year prior to Screening.
27. History of alcohol abuse within 3 months prior to Screening or consumes > 21 units per week for males and > 14 units per week for females. One unit of alcohol equals 12 oz (360 mL) beer, 1½ oz (45 mL) liquor, or 5 oz (150 mL) wine.
28. Subject has evidence of hepatorenal syndrome or creatinine clearance < 60 mL/minute as calculated by using the Cockcroft-Gault equation.
29. Subject has a current functioning organ transplant or is waiting for an organ transplant.
30. History of unstable diabetes mellitus as evidenced by hemoglobin A1c ≥ 9% at Screening.
31. Subjects with severe ascites and/or pleural effusion at Screening and Check-in.
32. Subject has had esophageal banding within 3 months prior to Check-in or required any other treatment for gastrointestinal bleeding within 6 months prior to Check-in.
33. Subjects with history of or current severe hepatic encephalopathy (Grade 2 or higher) within 3 months.
34. History or current diagnosis of uncontrolled or significant cardiac disease indicating significant risk of safety for participation in the study, including any of the following:

    1. Recent myocardial infarction (within 6 months of Check-in).
    2. New York Heart Association Class III or IV congestive heart failure.
    3. Unstable angina (within 6 months of Check-in).
    4. Clinically significant (symptomatic) cardiac arrhythmias (eg, sustained ventricular tachycardia, second- or third- degree atrioventricular block without a pacemaker).
    5. Uncontrolled hypertension.
35. Subjects with mild or moderate hepatic impairment ECG findings deemed clinically significant by the Investigator or Medical Monitor.
36. Subjects with any of the following laboratory results at Screening and Check-in:

    * Platelet count < 50,000/mm3
    * Hemoglobin <9 g/dL
37. Subjects with biliary liver cirrhosis or other causes of hepatic impairment not related to parenchymal disorder and/or disease of the liver, including hepatocellular carcinoma.
38. Subjects with history of portacaval shunt surgery, including transjugular intrahepatic portosystemic shunts.
39. Subjects with other causes of CP scores between 5 and 9 (inclusive) that are unrelated to hepatic impairment.

    Healthy Subjects with Normal Hepatic Function:
40. Use or intend to use any prescription medications/products other than hormone replacement therapy (HRT), and oral, implantable, transdermal, injectable, or intrauterine contraceptives within 30 days prior to dosing, unless deemed acceptable by the Investigator.
41. Use or intend to use any nonprescription medications/products including vitamins, minerals, and phytotherapeutic-/herbal-/plant-derived preparations within 7 days prior to Check-in, unless deemed acceptable by the Investigator. The occasional use of paracetamol/acetaminophen (not more than 2 g/day for up to 3 consecutive days) or other medication will be approved by Sponsor on a case-by-case basis.
42. History of drug abuse within 2 years prior to Screening.
43. History of alcohol abuse within 12 months prior to Screening or consumes > 21 units per week for males and > 14 units per week for females. One unit of alcohol equals 12 oz (360 mL) beer, 1½ oz (45 mL) liquor, or 5 oz (150 mL) wine.
44. Use of tobacco- or nicotine-containing products within 3 months prior to Check-in.
45. Positive urine cotinine test at Screening or Check-in.
46. Subject has creatinine clearance < 80 mL/minute as calculated by using the Cockcroft-Gault equation.
47. Use or intend to use slow-release medications/products considered to still be active within 30 days prior to IMP administration, unless deemed acceptable by the Investigator.
48. Subjects who tested positive at Screening for hepatitis C antibody indicating acute or chronic infection.
49. Significant history or clinical manifestation of any hepatic disease, as determined by lab abnormalities: aspartate aminotransferase, alanine aminotransferase, alkaline phosphatase, or alpha-fetoprotein > 1 × upper limit of normal or as deemed clinically significant by the Investigator.
50. Ventricular dysfunction or history of risk factors for Torsades de Pointes (eg, unexplained syncope, known long QT syndrome, heart failure, and cardiomyopathy). Subjects will be excluded if there is a family history of long QT syndrome. QTcF must not be > 450 ms for male subjects or > 470 ms for female subjects, or ECG findings deemed clinically significant by the Investigator or Medical Monitor.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2019-11-26 (Actual); Primary Completion 2020-03-20 (Actual); Study Completion 2020-03-20 (Actual)

PRIMARY OUTCOMES:
Cmax | Day 1 to Day 12
  Maximum observed concentration (KW-6356 and its major metabolite in plasma).
AUC0-t | Day 1 to Day 12
  AUC from time zero to the last quantifiable concentration (KW-6356 and its major metabolite in plasma).
AUC0-∞ | Day 1 to Day 12
  AUC from time zero to infinity (KW-6356 and its major metabolite in plasma).
tmax | Day 1 to Day 12
  Time of the maximum observed concentration (KW-6356 and its major metabolite in plasma).
t1/2 | Day 1 to Day 12
  Elimination half-life (KW-6356 in plasma).
CL/F | Day 1 to Day 12
  Apparent total clearance (KW-6356 in plasma).
Vz/F | Day 1 to Day 12
  Volume of distribution during terminal elimination phase (KW-6356 in plasma).

SECONDARY OUTCOMES:
Plasma protein binding of KW-6356 and its major metabolite | 1 hour after dosing Day 1, and 24 hours after dosing Day 2
Adverse Events | From screening through study completion, an average of 40 days.
  Number of subjects experiencing an adverse event related to treatment.
Clinical Laboratory Evaluations | From screening through study completion, an average of 40 days.
  Number of subjects with abnormal laboratory values that are related to treatment.
Vital signs | From screening through study completion, an average of 40 days.
  Number of subjects with abnormal vital signs that are related to treatment.
12-lead ECG | From screening through study completion, an average of 40 days.
  Number of subjects with abnormal ECG that are related to treatment.
Physical examination | From screening through study completion, an average of 40 days.
  Number of subjects with abnormal physical exam findings that are related to treatment.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Clinical Pharmacology of Miami, LLC, Miami, Florida
  - Orlando Clinical Research Center, Orlando, Florida
  - Pinnacle Clinical Research, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No